CLINICAL TRIAL: NCT03729258
Title: Comparison of the Efficacy and Safety of Immediate (b.i.d) and Modified (q.d.) Release Cefpodoxime Formulations in the Treatment of Acute Sinusitis: a Double-blind, Randomized, Phase III, Non-inferiority Study.
Brief Title: Efficacy and Safety of Modified Release Cefpodoxime Formulation in the Treatment of Acute Sinusitis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-04.15
Record Dates: First submitted 2018-10-22; First posted 2018-11-02 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Sinusitis; Sinusitis, Acute; Rhinosinusitis; Rhinosinusitis Acute; Sinus Infection
MeSH Terms: conditions — Sinusitis; Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefpodoxime 200 (b.i.d) (Experimental)
  Interventions: Drug: Infex 200 IR
- Cefpodoxime 400 (q.d) (Active Comparator)
  Interventions: Drug: Infex 400 MR

INTERVENTIONS:
Drug: Infex 400 MR — Infex (cefpodoxime) 400mg once a day (QD) for 10 days
  Arms: Cefpodoxime 400 (q.d)
Drug: Infex 200 IR — Infex (cefpodoxime) 200mg twice a day (BID) for 10 days
  Arms: Cefpodoxime 200 (b.i.d)

SUMMARY:
The aim of this study is to compare the efficacy and safety of cefpodoxime 200 mg immediate (b.i.d) and cefpodoxime 400 mg modified release (q.d) tablet formulations in the treatment of acute bacterial rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older patients who have acute bacterial rhinosinusitis sign and symptoms (i, ii, iii) according to IDSA Clinical Practice Guideline for Acute Bacterial Rhinosinusitis in Children and Adults: i. Onset with persistent symptoms or signs* compatible with acute rhinosinusitis, lasting for ≥ 10 days without any evidence of clinical improvement, ii. Onset with severe symptoms or signs of high fever > 39 and purulent nasal discharge or facial pain lasting for at least 3-4 consecutive days at the beginning of illness, iii. Onset with worsening symptoms or signs characterized by the new onset of fever, headache, or increase in nasal discharge that lasted 5-6 days and were initially improving.

   (*Major symptoms: Purulent anterior nasal discharge, Purulent or discolored posterior nasal discharge, Nasal congestion or obstruction, Facial congestion or fullness, Facial pain or pressure, d Hyposmia or anosmia. *Minor symptoms: Headache, Ear pain, pressure, or fullness, Halitosis, Dental pain, Cough, Fatigue)
2. Patients who are able to give culture sample from middle meatus (microorganisms to be teste: Streptococcus pneumoniae, Haemophilus influenzae [including beta-lactamase producing strains], Streptococcus pyogenes and Moraxella catarrhalis [including beta-lactamase producing strains]).
3. Patients who are able to use oral drugs,
4. If patient is a women of childbearing age; female patients who applies appropriate birth control,
5. Patients who have ability to communicate with investigators,
6. Patients who commits to adhere to the study protocol,
7. Patients who sign informed consent form.

Exclusion Criteria:

1. Patients who have hypersensitivity to beta-lactam antibiotics, penicillin and cefpodoxime,
2. Patients who hypersensitivity to peanut and soy,
3. Patients who have kidney or liver deficiency,
4. Patients who have history of more than 2 bacterial sinusitis episode within last 12 months,
5. Patients who have chronic sinusitis,
6. Patients who have history of head and neck surgery and/or severe sinusitis complication (brain abscess or venous thrombosis),
7. Patients who are hospitalized within 4 weeks prior to the start of study,
8. Patients who have immunodeficiency (i.e; HIV, corticosteroid use, immunosuppressive use),
9. Patients who used antibiotics within 30 days prior to the start of study,
10. Patients who need to use of antibiotics other than investigational drugs for concomitant disease,
11. Patients who used aluminium and magnesium containing anti-acids, probenecid and iron containing drugs within 2 weeks prior to the start of study,
12. Pregnant and lactating female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of formulations on acute sinusitis symptoms | 10 days
  Change in acute sinusitis sign and symptoms at the end of treatment compared to baseline.
  The outcome will be assessed by Sino-nasal Outcome Tests SNOT-22 and SNOT-16.
  * SNOT-16 is recommended symptom questionnarie for acute rhinonusitis but Turkish validation is not existed. Therefore SNOT-22 is also added as a symptom questionnarie since Turkish Validation is available.
Effect of formulations on quality of life scale | 10 days
  Quality of Life: Increase or decrease in quality of life. The outcome will be assessed by Short Form Health Survey (SF-12).
Rate of microbiological response at the end of treatment | 10 days
  Patients will be given sample from middle meatus.
  The outcome will be assessed according to microbiologic response:
  Eradication: The absence of pathogen(s) at the end of treatment. Persistance: The same concentration of the pathogen(s) in culture after the end of treatment.
  Superinfection: Detection of bacterial of fungal pathogens during or after treatment,

SECONDARY OUTCOMES:
Evaluation of the safety of investigational products | 10 days
  Number of Adverse Events That Are Related to Treatments and Participants with Abnormal Laboratory Values (hemogram, sedimentation, CRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided